CLINICAL TRIAL: NCT03028116
Title: A Randomized, Blinded, Placebo-controlled Study of Phase I Allantoic Split Inactivated Seasonal Influenza Vaccine in Healthy Adults
Brief Title: Reactogenicity, Safety and Immunogenicity Study of a Allantoic Split Inactivated Seasonal Influenza Vaccine
Acronym: VSI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Research Institute for Biological Safety Problems (Other Government)
Collaborators: Asfendiyarov Kazakh National Medical University (Other); Research Institute of Influenza, Russia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VSI-I-01/2016
Record Dates: First submitted 2017-01-04; First posted 2017-01-23 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2016-12

CONDITIONS: Influenza, Human
Keywords: vaccine; 1 phase; safety
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allantoic split inactivated seasonal influenza vaccine (Active Comparator): Allantoic split inactivated seasonal influenza vaccine
  Interventions: Biological: influenza vaccine
- Placebo (Placebo Comparator): Water for Injection
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: influenza vaccine — A allantoic split inactivated seasonal influenza vaccine has been prepared on eggs and is made from inactivated parts of the following influenza virus strains:
  NIBRG-121xp (A/California/7/2009 (H1N1)v and А/PR/8/34 (H1N1)), NYMC X-217 (A/Victoria/361/2011(H3N2) and А/PR/8/34 (H1N1)), NYMC BX-49 (B/Texas/06/2011 (Yamagata lineage) - like High Yield Reassortant (1:1:6) With B/Lee/40 NP, B/Panama/45/90 NS genes).
  Arms: Allantoic split inactivated seasonal influenza vaccine
Biological: Placebo — water for injection
  Arms: Placebo

SUMMARY:
The study is a single centre, phase I, double-blind, randomized, placebo-controlled trial that explored the safety and immunogenicity of single dose a allantoic split inactivated seasonal influenza vaccine in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers of both sexes aged 18-60 years.
* Persons seronegative against A/H1N1 influenza virus, A/H3N2 and type B (with antibody titers ≤1: 10, according to hemagglutination-inhibition (HI) assay to determine).
* Literate and willing to provide written informed consent.
* A signed informed consent.

Exclusion Criteria:

* Available in anamnaze volunteer at any allergic reactions.
* Allergic reactions to chicken proteins, or any preceding vaccination.
* Acute illness with a fever (37.0 C).
* Vaccination against influenza in the 2012/2013 season.
* Seropositive volunteers against A/H1N1 influenza virus, A/H3N2 and type B (with antibody titers greater than 1:10 according HI).
* Current or recent (within two weeks of enrollment) acute respiratory illness with or without fever.
* Hypersensitivity after previous administration of any vaccine.
* History of chronic alcohol abuse and/or illegal drug use.
* Any clinically significant abnormal laboratory finding.
* A positive pregnancy test for all women of childbearing potential.
* Administration of immunosuppressive drugs or other immune modifying drugs within 4 weeks prior to study enrollment.
* Acute or chronic clinically significant pulmonary disease, cardiovascular disease, gastrointestinal disease, liver disease, neurological illness, liver disease, blood disease, skin disorder, endocrine disorder, neurological illness and psychiatric disorder as determined by medical history, physical examination or clinical laboratory screening tests, which in the opinion of the investigator, might interfere with the study objectives.
* History of leukemia or any other blood or solid organ cancer.
* Seropositive for HIV, hepatitis B surface antigen and/or hepatitis C antibodies.
* Receipt of antivirals, antibiotics, immunoglobulins or other blood products within 4 weeks prior to study enrollment or planned receipt of such products during the period of subject participation in the study.
* Participation in another clinical trial within the previous three months or planned enrollment in such a trial during the period of this study.
* Subjects who are, in the opinion of the investigator, at significantly increased risk of non-cooperation with requirements of the study protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2016-05; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Solicited Local and Systemic Adverse Events (AEs) | Two hours
  Participants recorded solicited injection site and systemic adverse events in a Subject Diary. Solicited Locals AEs were: Injection Site Pain, Injection Site Redness, Injection Site Swelling, Injection Site Induration and Injection Site Ecchymosis. Solicited Systemic AEs were: Pyrexia, Malaise, Chills, Fatigue, Headache, Sweaty, Myalgia, Arthralgia, Nausea and Vomiting.
Percentage of Participants Reporting One or More Treatment-emergent Adverse Events (TEAE) | Greater than 2 hours after administration of any dose of vaccine or placebo through 7 days following any dose
  Adverse events are defined as unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product, regardless of relationship to the medicinal product. TEAE is defined as an adverse event with an onset that occurs after receiving study drug.
Percentage of Participants With Abnormal Safety Laboratory Tests at Least Once Post Dose Reported as AEs | Greater than 2 hours after administration of any dose of vaccine or placebo through 7 days
  The percentage of participants with any abnormal standard safety laboratory values (Chemistry, Hematology and Urinalysis) collected throughout the study reported as AEs.
Serious adverse events (SAEs), including abnormal laboratory findings | Three weeks of receipt
  Serious adverse events (SAEs) are medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.

SECONDARY OUTCOMES:
Geometric Mean Fold Increase in HI Antibody Titer | Change from Baseline HI Antibody Titer at 21 days
  Geometric mean fold increase in HI antibody titer for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after vaccination, as compared with Baseline.
Seroconversion Rate of Hemagglutination Inhibition (HI) Antibody Titer | Change from Baseline HI Antibody Titer at 21 days
  Seroconversion rate was measured by hemagglutination inhibition (HI) antibody titer for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after vaccination. Seroconversion rate was defined as the percentage of participants achieving a minimal 4-fold increase from the Baseline HI antibody titer in participants with a Baseline titer ≥10, or achieving an HI antibody titer of ≥40 in participants with a Baseline titer <10.
Seroprotection Rate of HI Antibody Titer | Change from Baseline HI Antibody Titer at 21 days
  Seroprotection rate, defined as the percentage of participants with HI antibody titer of ≥40, was measured by HI antibody titer for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after vaccination. Day 1 data is reported for reference.

CONTACTS AND LOCATIONS:
Locations (1):
- Kazakh National Medical University, Almaty, Almaty, Kazakhstan

IPD SHARING:
Plan to Share IPD: Undecided